CLINICAL TRIAL: NCT00790803
Title: Vascular Endothelial Growth Factor (VEGF)Blockade With Intravitreal Pegaptnib in Non-Infectious Uveitic Cystoid Macular Edema (CME)
Brief Title: Pegaptanib Therapy in Non-Infectious Uveitic Cystoid Macular Edema
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University (Other)
Responsible Party: Sponsor
Organization: Wake Forest University Health Sciences (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 4499 Pegaptanib in uveitis
Record Dates: First submitted 2008-11-12; First posted 2008-11-14 (Estimated); Results first posted 2013-09-26 (Estimated); Last update posted 2022-03-15 (Actual); Status verified 2017-02

CONDITIONS: Uveitis; Cystoid Macular Edema
Keywords: uveitis; cystoid macular edema
MeSH Terms: conditions — Uveitis; Macular Edema | interventions — pegaptanib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Pegaptanib (Macugen) (Other): Open label, non randomized, interventional controlled injection of 0.3mg of Pegaptanib (Macugen) every 6weeks with max of 5 injections over 30weeks.
  Interventions: Drug: Pegaptanib

INTERVENTIONS:
Drug: Pegaptanib — Five patients will receive intravitreous injections of Macugen 0.3 mg every 6 weeks as needed for a total of no more than five.
  Other Names: Macugen

SUMMARY:
According to a recent estimate more than 280,000 people in the United States are affected by uveitis each year. This report, also estimated that uveitis is the reason for 30,000 new cases of blindness/year and up to 10 percent of all cases of blindness. The purpose of this trial is to determine the effectiveness of VEGF blockade with intravitreal pegaptanib in patients with uveitic CME.

DETAILED DESCRIPTION:
1. Cystoid macular edema is a common complication of uveitic intraocular inflammatory diseases and is characterized by intraretinal edema involving the outer plexiform layer. Intraocular inflammation or uveitis may be associated with non infectious or infectious etiologies. The early symptoms of CME include a decrease or blurry central vision. With long standing CME there is a substantial risk of photoreceptor degeneration and ensuing long term decrease in the quality and level of visual acuity (VA). Furthermore it has been shown that in patients with uveitis, the morphologic features of macular edema and macular thickness correlated with final VA. Current therapeutic interventions have had at best modest results in patients with CME who have had decreased VA. This may the case with systemic interventions also.
2. Vascular endothelial growth factor is a very strong inducer of blood vessel permeability and has been linked to the ocular manifestations of uveitis including CME by experienced researchers both in experimental and clinical settings. In animal tests, VEGF has been shown to be 50,000 times more potent than histamine, the molecule commonly associated with blood vessel leakage related to allergies. Also in animal tests, it has been shown that VEGF is required for the blood vessel permeability associated with neovascular AMD and diabetic retinopathy that have been shown to have an inflammatory component. In addition to its anti-angiogenic property of inhibiting abnormal blood vessel growth, pegaptanib has been shown in animal tests to inhibit blood vessels from leaking into the retina. Uveitis has been shown to be associated with ocular neovascularization both clinically and well as in the clinical studies. Thus, by preventing blood vessel leakage as well as abnormal blood vessel growth pegaptanib may be a viable approach for the treatment of CME. Although pegaptanib use has been associated with mild transient anterior segment inflammation CME itself has not been linked to its use. Besides, pegaptanib has been demonstrated to effect a sustainable decrease the macular edema in maculopathies, both age related and diabetic.
3. There is currently a need for considering alternative forms of local (ocular) therapy for CME to triamcinolone (sub tenon and intraocular). The serious adverse effects with intraocular corticosteroid use are well documented and include cataracts (nuclear and subcapsular), glaucoma, endophthalmitis (may be significantly higher than pegaptanib in patients who are treated exactly as per protocol) as well as sterile inflammatory reactions.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female adults (>18 years of age) with non infectious uveitis.
2. Demonstrable (FA and/or OCT) bilateral or unilateral CME associated with uveitis of greater than 3 months but less than 1 years duration that is documented by two independent qualified observers.
3. Best corrected VA between 20/40 and 20/200 as measured by the ETDRS chart attributable to CME in the study eye.
4. Patients may be receiving systemic therapy for the treatment of their intraocular inflammation or cystoid macular edema, or may have been treated for the cystoid macular edema in the past.
5. Anterior chamber inflammation equal to or greater than 1+ and vitreous inflammation equal to or greater than 1+ cell and 1+ haze as per the 'Standardization of Uveitis' working group definition.
6. Females of child bearing potential must agree to utilize effective contraception during the study and two months after the last dose of study medication.
7. Male study patients will agree to use effective contraception.
8. Ability to give informed consent.

Exclusion Criteria:

1. Allergy to pegaptanib or any of its components
2. Diabetic retinopathy, macular degeneration or any other ocular condition affecting the study eye that may cause vision loss or in the opinion of the study investigator would interfere with the evaluation of the efficacy of Macugen for the treatment of uveitis associated CME.
3. Refusal to try the therapeutic alternative pegaptanib
4. Lack of understanding of the consent or protocol
5. Suspicion/proved history or current diagnosis, (clinical or otherwise) of infectious uveitis.
6. Need for intraocular surgery within 30 weeks of study duration.
7. Periocular steroids to the study eye less than 6 weeks prior to study enrollment
8. History of any prior intravitreal injections in study eye
9. Systemic immunomodulatory agent(s) added or increased in dosage (>20%) within the last two months prior to study enrollment, or potential need for any increase during the study.
10. Requirement for systemic corticosteroids in the equivalent of oral prednisone > 30mg/day
11. Topical prostaglandin analog use
12. Severe debilitating disease or medical problems that make consistent follow-up over the treatment period unlikely (e.g. liver impairment, stroke, severe myocardial infarction, terminal cancer).
13. History of hypersensitivity to fluorescein or multiple drug allergies that may increase the chance of a drug reaction to Macugen.
14. Unclear media that precludes assessment of cystoid macular edema in eligible eye(s), such as a cataract or vitreal opacity.
15. Evidence of a macular hole in the study eye.
16. Prior or current retinal detachment in the study eye.
17. Concurrent treatment with any new investigational drug.
18. Pregnant or lactating women (Pregnant and lactating women are excluded since pregnancy may have some effect on CME).
19. Inability to comply with the study requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2009-03; Primary Completion 2011-11 (Actual); Study Completion 2012-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shree Kurup, MD, Principal Investigator — Wake Forest University Eye Center
Locations (1):
- Wake Forest University Eye Center, Winston-Salem, North Carolina, United States

REFERENCES:
- [Background] Gritz DC, Wong IG. Incidence and prevalence of uveitis in Northern California; the Northern California Epidemiology of Uveitis Study. Ophthalmology. 2004 Mar;111(3):491-500; discussion 500. doi: 10.1016/j.ophtha.2003.06.014. PMID 15019324
- [Background] Okhravi N, Lightman S. Cystoid macular edema in uveitis. Ocul Immunol Inflamm. 2003 Mar;11(1):29-38. doi: 10.1076/ocii.11.1.29.15582. PMID 12854025
- [Background] Kurup SK, Chan CC. Immunotherapeutic approaches in ocular inflammatory diseases. Arch Immunol Ther Exp (Warsz). 2005 Nov-Dec;53(6):484-96. PMID 16407781
- [Background] Vinores SA, Chan CC, Vinores MA, Matteson DM, Chen YS, Klein DA, Shi A, Ozaki H, Campochiaro PA. Increased vascular endothelial growth factor (VEGF) and transforming growth factor beta (TGFbeta) in experimental autoimmune uveoretinitis: upregulation of VEGF without neovascularization. J Neuroimmunol. 1998 Aug 14;89(1-2):43-50. doi: 10.1016/s0165-5728(98)00075-7. PMID 9726824
- [Background] Kurup SK, Chan CC. Mycobacterium-related ocular inflammatory disease: diagnosis and management. Ann Acad Med Singap. 2006 Mar;35(3):203-9. PMID 16625271
- [Background] Rothova A. Medical treatment of cystoid macular edema. Ocul Immunol Inflamm. 2002 Dec;10(4):239-46. doi: 10.1076/ocii.10.4.239.15589. PMID 12854032
- [Background] Markomichelakis NN, Halkiadakis I, Pantelia E, Peponis V, Patelis A, Theodossiadis P, Theodossiadis G. Patterns of macular edema in patients with uveitis: qualitative and quantitative assessment using optical coherence tomography. Ophthalmology. 2004 May;111(5):946-53. doi: 10.1016/j.ophtha.2003.08.037. PMID 15121373
- [Background] Fine HF, Baffi J, Reed GF, Csaky KG, Nussenblatt RB. Aqueous humor and plasma vascular endothelial growth factor in uveitis-associated cystoid macular edema. Am J Ophthalmol. 2001 Nov;132(5):794-6. doi: 10.1016/s0002-9394(01)01103-5. PMID 11704050
- [Background] Krzystolik MG, Filippopoulos T, Ducharme JF, Loewenstein JI. Pegaptanib as an adjunctive treatment for complicated neovascular diabetic retinopathy. Arch Ophthalmol. 2006 Jun;124(6):920-1. doi: 10.1001/archopht.124.6.920. No abstract available. PMID 16769855
- [Background] Kourlas H, Schiller DS. Pegaptanib sodium for the treatment of neovascular age-related macular degeneration: a review. Clin Ther. 2006 Jan;28(1):36-44. doi: 10.1016/j.clinthera.2006.01.009. PMID 16490578
- [Background] Cunningham ET Jr, Adamis AP, Altaweel M, Aiello LP, Bressler NM, D'Amico DJ, Goldbaum M, Guyer DR, Katz B, Patel M, Schwartz SD; Macugen Diabetic Retinopathy Study Group. A phase II randomized double-masked trial of pegaptanib, an anti-vascular endothelial growth factor aptamer, for diabetic macular edema. Ophthalmology. 2005 Oct;112(10):1747-57. doi: 10.1016/j.ophtha.2005.06.007. PMID 16154196
- [Background] VEGF Inhibition Study in Ocular Neovascularization (V.I.S.I.O.N.) Clinical Trial Group; D'Amico DJ, Masonson HN, Patel M, Adamis AP, Cunningham ET Jr, Guyer DR, Katz B. Pegaptanib sodium for neovascular age-related macular degeneration: two-year safety results of the two prospective, multicenter, controlled clinical trials. Ophthalmology. 2006 Jun;113(6):992-1001.e6. doi: 10.1016/j.ophtha.2006.02.027. Epub 2006 Apr 27. PMID 16647134
- [Background] Amato JE, Lee DH, Santos BA, Akduman L. Steroid hypopyon following intravitreal triamcinolone acetonide injection in a pseudophakic patient. Ocul Immunol Inflamm. 2005 Apr-Jun;13(2-3):245-7. doi: 10.1080/09273940590928562. PMID 16019686
- [Background] Konstantopoulos A, Williams CP, Newsom RS, Luff AJ. Ocular morbidity associated with intravitreal triamcinolone acetonide. Eye (Lond). 2007 Mar;21(3):317-20. doi: 10.1038/sj.eye.6702416. Epub 2006 May 19. PMID 16710433

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Five patients with non-infectious uveitis, ongoing for greater than three months but less than twelve months with associated CME. Patients were identified in the PI's regular medical clinic and received five intravitreal pegaptanib doses over the course of thirty weeks.
Pre-assignment Details: Five consecutive adult patients with non-infectious uveitis associated CME were chosen for this study. Only patients with a baseline best corrected VA between 20/40 and 20/200, attributable to CME, were selected for the study. In qualified patients with bilateral disease, the eye with the worse visual acuity was selected for the study eye.
Groups:
- Macugen: Single arm pilot trial
  Pegaptanib (Macugen) : Five patients will receive intravitreous injections of Macugen 0.3 mg every 6 weeks as needed for a total of no more than five.
Period: Overall Study
Arm/Group | Macugen
Started | 5
Completed | 5
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Macugen
Number analyzed (Participants) | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 4
  >=65 years | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.8 (19.05781)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 1
Region of Enrollment [Number; unit: participants]
  United States | 5

OUTCOME MEASURES:

1. Primary Outcome: Improvement in VA ETDRS >/= 15 Letters
Description: The primary outcome was an improvement in VA greater than or equal to fifteen letters on the EDTRS chart.
Time Frame: 32 weeks
Population: Five consecutive adult patients with non-infectious uveitis associated CME were chosen from the PI's regular medical clinic. Patients demonstrated, on fluorescein angiogram and/or optical tomography, bilateral or unilateral CME with non-infectious uveitis for greater than three months, but less than twelve.
Measure: Number; unit: participants
Arm/Group | Macugen
Number analyzed (Participants) | 5
participants | 1

2. Secondary Outcome: Proportion of Patients Experiencing > 0 Letter Vision Gain and a < 15 Loss
Description: Patients best corrected visual acuity was measured at each visit to monitor gain or loss of letters on the EDTRS chart.
Time Frame: 32 weeks
Measure: Number; unit: paticipants
Arm/Group | Macugen
Number analyzed (Participants) | 5
paticipants | 5

3. Secondary Outcome: Decrease in CME as Evidenced by Imaging (Fluorescein Angiography and 50 Micron Change in OCT)
Description: Patients retinal thickness was measured at each visit bu imaging to monitor increase or decrease in thickness.
Time Frame: 32 weeks
Measure: Number; unit: participants
Arm/Group | Macugen
Number analyzed (Participants) | 5
participants | 2

4. Secondary Outcome: A Decrease in Anterior Chamber Cells or Vitreous Cells or Haze in Injected Eye
Description: The degree of cell and flare was recorded at each visit during the course of the trial in the injected eye.
  In uveitis, severely inflamed vessels leak protein which clouds the normally clear aqueous. This looks hazy with the slit lamp. If severe, it disperses the light beam, causing flare.
  White or red blood cells may be observed: the presence of inflammatory cells in the anterior chamber suggests inflammation of the iris and ciliary body.
  Blood cells: grading of blood cells in the anterior chamber is as follows:
  * 0 - None.
  * 1+ - faint (barely detectable).
  * 2+ - moderate (clear iris and lens details).
  * 3+ - moderate (hazy iris and lens details).
  * 4+ - intense (fibrin deposits, coagulated aqueous).
Time Frame: 32 weeks
Measure: Number; unit: participants
Arm/Group | Macugen
Number analyzed (Participants) | 5
participants | 0

5. Secondary Outcome: Change in Immunomodulatory Medications (Topical, Periocular or Systemic) After the Initiation of Macugen Therapy
Description: No changes were to be made in immunodulatory medications of the patients unless needed for safety after in initiation of Macugen therapy.
Time Frame: 32 weeks
Measure: Number; unit: participants
Arm/Group | Macugen
Number analyzed (Participants) | 5
participants | 0

ADVERSE EVENTS:
Arm/Group | Macugen
Serious Adverse Events (participants affected / at risk) | 0/5
Other Adverse Events (participants affected / at risk) | 0/5

LIMITATIONS AND CAVEATS:
Implementing screening protocols to catch less progressed CME cases could improve outcomes.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes